CLINICAL TRIAL: NCT05401162
Title: Conventional Dose Chemotherapy for Ovarian Cancer Supported by Autologous Haematopoietic Stem Cell Transfusion
Brief Title: Chemotherapy Supported by Autologous Hematopoietic Stem Cells
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG0203
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Conventional chemotherapy; blood stem cells; autologous blood transfusion
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Blood Transfusion, Autologous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): transfusion of autologous blood containing haematopoietic stem cells after conventional chemotherapy
  Interventions: Other: Autologous blood transfusion with haematopoietic stem cells
- Control group (No Intervention): enrolled ovarian cancer patients receive conventional chemotherapy

INTERVENTIONS:
Other: Autologous blood transfusion with haematopoietic stem cells — Transfusion of autologous blood containing haematopoietic stem cells for haematopoietic reconstruction after chemotherapy.Blood tests were performed weekly, if the patient's neutrophils were less than 1.0 × 109 / L during chemotherapy, G-CSF was given as a remedial treatment. If fever occurs, antibiotics were given promptly.Monitor peripheral blood after transfusion. If peripheral blood leukocyte count does not reach 1.0 x 109/L, administer G-CSF 150 μg subcutaneously daily until peripheral blood leukocyte count reaches 1.0 x 109/L.Patients were tested monthly for peripheral blood cells for 6 months after the end of treatment.
  Arms: Experimental group

SUMMARY:
The aim of this project is to use autologous haematopoietic stem cell transfusion support to promote the reconstruction of haematopoietic function after chemotherapy for ovarian cancer. To explore the impact of stored haematopoietic stem cell support therapy on bone marrow protection after conventional chemotherapy for ovarian cancer in order to facilitate its clinical application.

DETAILED DESCRIPTION:
Study design:In this prospective, single-center,non-randomised controlled study, patients with ovarian cancer were divided into two groups. The patients in the experimental group received autologous blood transfusion containing hematopoietic stem cells 1 day after conventional chemotherapy, while the control group only received conventional chemotherapy.

Case selection: Patients with primary ovarian cancer,ovarian cancer confirmed by histopathology, and three weeks of platinum-containing regimen chemotherapy.

Primary end point: 1)incidence and duration of grade 3/4 neutropenia in patients;2)hematopoietic reconstitution time in patients. Secondary endpoints: 1)the rate of reduction in chemotherapy dose and postponement of the course for chemotherapy;2) Incidence of febrile neutropenia (FN);3)Safety of hematopoietic stem cell reinfusion therapy (adverse events).

Safety assessment: laboratory safety testing, including platelet count,white blood cell and hemoglobin. Evaluation of adverse events: infection, neutropenic fever, hypocalcemia,anemia and thrombocytopenia,bone pain, etc.

ELIGIBILITY:
Inclusion Criteria:

1）18-60 years old; 2)there are chemotherapy indicators for ovarian cancer;3)ovarian cancer diagnosed by histopathology;4)recurrent and metastatic ovarian cancer;5)the Eastern Cooperative Oncology Group (ECOG) performance status score≤1;6)the expected survival time was more than 3 months; 7)pre-menopausal women (post-menopausal women must have been postmenopausal for at least 12 months to be considered infertile), and the serum pregnancy test results are negative;8)all patients must agree to take effective contraceptive measures during the study period and within 6 months after stopping treatment;9)the subjects voluntarily participate in this clinical trial sign an informed consent form and are able to complete the study procedures and follow-up examinations;10)bone marrow function is good,ability to perform stem cell mobilisation and collection.

Exclusion Criteria:

1) patients with bone marrow disease;2)central nervous system or soft meningeal or bone or bone marrow metastases confirmed by imaging or pathology;3)patient has severe cardiac insufficiency;4)previous history of allogeneic stem cell transplantation or organ transplantation;5)patients with active bleeding and autoimmune thrombocytopenic purpura;6)patients with chemotherapy contraindications;7)positive for human immunodeficiency virus (HIV);8)acute or chronic active hepatitis B or hepatitis C infection.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 3-4 neutropenia | 8 months
  Incidence of Grade 3-4 neutropenia
Time to reconstruct haematopoietic function | 8 months
  Time to reconstruct haematopoietic function
Incidence of febrile neutropenia (FN) | 8 months
  Incidence of febrile neutropenia (FN)

SECONDARY OUTCOMES:
the rate of postponement of the course for chemotherapy | 8 months
  the rate of postponement of the course for chemotherapy
reduction in chemotherapy dose | 6 months
  reduction in chemotherapy dose
Safety of hematopoietic stem cell reinfusion therapy | 3 months
  Safety of hematopoietic stem cell reinfusion therapy(adverse events)

CONTACTS AND LOCATIONS:
Overall Officials: Dongling Zou, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weycker D, Bensink M, Wu H, Doroff R, Chandler D. Risk of chemotherapy-induced febrile neutropenia with early discontinuation of pegfilgrastim prophylaxis based on real-world data from 2010 to 2015. Curr Med Res Opin. 2017 Dec;33(12):2115-2120. doi: 10.1080/03007995.2017.1386638. Epub 2017 Oct 16. PMID 28958156
- [Background] Cooper KL, Madan J, Whyte S, Stevenson MD, Akehurst RL. Granulocyte colony-stimulating factors for febrile neutropenia prophylaxis following chemotherapy: systematic review and meta-analysis. BMC Cancer. 2011 Sep 23;11:404. doi: 10.1186/1471-2407-11-404. PMID 21943360
- [Background] Magagnoli M, Masci G, Castagna L, Rimassa L, Bramanti S, Santoro A. Intermediate-dose melphalan with stem-cell support in platinum-refractory ovarian cancer. Bone Marrow Transplant. 2004 Jun;33(12):1261-2. doi: 10.1038/sj.bmt.1704527. No abstract available. PMID 15107813
- [Background] Ikeba K, Okubo M, Takeda S, Kinoshita K, Maeda H. Five-year results of cyclic semi-high dose neoadjuvant chemotherapy supported by autologous peripheral blood stem-cell transplantation in patients with advanced ovarian cancer. Int J Clin Oncol. 2004 Apr;9(2):113-9. doi: 10.1007/s10147-003-0377-x. PMID 15108043
- [Background] Aghajanian C, Fennelly D, Shapiro F, Waltzman R, Almadrones L, O'Flaherty C, O'Conner K, Venkatraman E, Barakat R, Curtin J, Brown C, Reich L, Wuest D, Norton L, Hoskins W, Spriggs DR. Phase II study of "dose-dense" high-dose chemotherapy treatment with peripheral-blood progenitor-cell support as primary treatment for patients with advanced ovarian cancer. J Clin Oncol. 1998 May;16(5):1852-60. doi: 10.1200/JCO.1998.16.5.1852. PMID 9586901
- [Background] Papadimitriou C, Dafni U, Anagnostopoulos A, Vlachos G, Voulgaris Z, Rodolakis A, Aravantinos G, Bamias A, Bozas G, Kiosses E, Gourgoulis GM, Efstathiou E, Dimopoulos MA. High-dose melphalan and autologous stem cell transplantation as consolidation treatment in patients with chemosensitive ovarian cancer: results of a single-institution randomized trial. Bone Marrow Transplant. 2008 Mar;41(6):547-54. doi: 10.1038/sj.bmt.1705925. Epub 2007 Nov 19. PMID 18026149
- [Background] Donato ML, Gershenson D, Ippoliti C, Wharton JT, Bast RC Jr, Aleman A, Anderlini P, Gajewski JG, Giralt S, Molldrem J, Ueno N, Lauppe J, Korbling M, Boyer J, Bodurka-Bevers D, Bevers M, Burke T, Freedman R, Levenback C, Wolf J, Champlin RE. High-dose ifosfamide and etoposide with filgrastim for stem cell mobilization in patients with advanced ovarian cancer. Bone Marrow Transplant. 2000 Jun;25(11):1137-40. doi: 10.1038/sj.bmt.1702421. PMID 10849525